CLINICAL TRIAL: NCT02930252
Title: Covered Versus Uncovered Self-conformable Metal Stent for Palliation of Primary Malignant Extra-hepatic Biliary Strictures: a Randomized Multicenter Study
Brief Title: Covered Versus Uncovered SEMS for Palliation of Malignant Biliary Strictures.
Acronym: SEMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL 1 Imperiese (Other)
Collaborators: Ospedali Riuniti Marche Nord, Pesaro, Italy (Unknown); NOCSAE Hospital, Modena, Italy (Unknown); University of Siena, Italy (Unknown); Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, MASSIMO CONIO, MD, Director of Gastroenterology Department, General Hospital Sanremo, Italy, Azienda USL 1 Imperiese
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 055REG2013
Record Dates: First submitted 2016-10-07; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Biliary Cancer
Keywords: Self-expandable metal stent; strictures; biliary
MeSH Terms: conditions — Biliary Tract Neoplasms; Constriction, Pathologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Niti-S Biliary ComVi Stent (Experimental): Device:
  Niti-S Biliary ComVi Stent is a hollow cylindrical stent fabricated by knitting first and second super-elastic shape memory alloy wires to make a net-like structure. A plurality of interlocked points allow each of the inside and outside stent bodies to contract and expand in the longitudinal direction and to apply a force against the longitudinal contraction. A hollow polytetrafluoroethylene (PTFE) membrane tube is closely fitted between the inside and outside stent bodies, with each of overlapped ends of the PTFE membrane tube and the inside and outside stent bodies integrated into a single structure.
  Interventions: Device: Niti-S Biliary ComVi Stent
- Niti-S Stent (D-type) (Active Comparator): Device:
  The Niti-S Stent (D-type) maintains a desired bent shape corresponding to the specific target lesion. It is comprised of a hollow cylindrical stent body fabricated by knitting first and second super-elastic shape memory alloy wires to make a net-like structure with a plurality of interlocked points capable of allowing the stent body to contract and expand in the longitudinal direction and to apply a force against the longitudinal contraction of the stent body.
  The wires are made of a shape memory alloy through a process of shaping the alloy then heat-treating the wires to allow restoration of the original shape at a predetermined temperature.
  Interventions: Device: Niti-S stent (D type)

INTERVENTIONS:
Device: Niti-S Biliary ComVi Stent — Endoscopic placement of biliary fully covered metal stents
  Other Names: Fully Covered biliary stent
  Arms: Niti-S Biliary ComVi Stent
Device: Niti-S stent (D type) — Endoscopic placement of biliary uncovered metal stent
  Other Names: Uncovered biliary stent
  Arms: Niti-S Stent (D-type)

SUMMARY:
The purpose of this study is to compare the duration of stent patency of a covered vs. an uncovered biliary self-expandable metal stents (SEMS) placed to relieve biliary obstruction in patients with inoperable extrahepatic malignant biliary obstruction.

DETAILED DESCRIPTION:
Cancer of the pancreas, gallbladder, or bile ducts is the most common cause of malignant obstruction of the biliary tree. Patients who have unresectable tumors have a dismal prognosis in terms of survival and quality of life. In these cases 5-year survival is less than 2% and palliation, such as the establishment of a biliary drainage, is the only treatment available. Two types of stents are routinely used: plastic stents (PS) and self-expandable metal stents (SEMS). The first generation SEMS are uncovered and recurrent obstruction, most frequently caused by tumor ingrowth through the metal mesh, is seen in 16-46%. Recently, covered SEMS have been introduced to prevent tumor ingrowth. Covered SEMS are associated with stent occlusion in 14% of patients. As can be expected, the most frequent cause of stent obstruction in these patients is sludge formation. Stent migration, and cholecystitis and pancreatitis caused by obstruction of the cystic duct and pancreatic duct, respectively, have been suggested to occur more frequently with covered SEMS. To date, however, one randomized trial and three comparative studies compared covered with uncovered SEMS, have found only a non statistically significant trend towards more frequent occurrence of these complications.

From these initial studies comparing uncovered to covered SEMS, it suggested that stent patency may be longer with covered SEMS. However, supporting evidence for the superior efficacy of covered SEMS is lacking. In addition, the issue of safety of covered SEMS, as well as the real world effectiveness of the self conformable SEMS, warrant further investigation.

In this study, the Investigators will include patients with symptoms (jaundice, cholangitis) due to malignant extrahepatic biliary tree obstruction (pancreatic cancer, cholangiocarcinoma, gallbladder cancer, or metastatic lymphadenopathy) who are not candidates for surgical cure either because the tumor is inoperable or because of the patient's poor medical condition due to comorbidities and/or advanced age.

Patients with extrahepatic malignancy in whom a diagnostic work up is still ongoing to establish the possibility of performing a curative approach will not be immediately enrolled. Patients who have been previously treated with a plastic stent will be eligible if the plastic stent was placed within the 4 weeks prior to enrolment in this study.

The purpose of this study is to compare the duration of stent patency of a covered vs. an uncovered biliary self-expandable metal stents (SEMS) placed to relieve biliary obstruction in patients with inoperable extrahepatic malignant biliary obstruction.

1. Primary Aim: To compare the duration of stent patency of a covered vs. an uncovered biliary SEMS placed to relieve biliary obstruction in patients with inoperable extrahepatic malignant biliary obstruction.

Secondary Aims:

In patients with inoperable extrahepatic malignant biliary obstruction managed with SEMS:

1. To evaluate complication rates of covered vs. uncovered biliary SEMS
2. To evaluate the quality of life before and after intervention with covered vs. uncovered biliary SEMS
3. To evaluate the survival of patients treated with covered vs. uncovered biliary SEMS
4. To evaluate the cost-effectiveness of covered and uncovered biliary SEMS
5. To determine the predictors of survival in patients in patients with inoperable extrahepatic malignant biliary obstruction managed with SEMS.

1.1 Primary endpoints

* Normalization of the bilirubin level and other cholestasis parameters
* Absence of clinically significant stent occlusion or migration prior to death of patients (minimum follow-up: 4 months) as defined below Clinically Significant Occlusion

It will be defined as an occurrence of the following items:

* The development of clinical symptoms of biliary obstruction such as cholangitis, accompanied by jaundice and fever requiring antibiotic treatment, and pruritis
* Laboratory evidence of cholestasis, including elevation of conjugated bilirubin (≥ 30% increase in bilirubin), alkaline phosphatase (ALP), aspartate aminotransferase (AST) and alanine transaminase (ALT) following stent placement
* Imaging findings consistent with biliary obstruction Initial stent failure: if normalization of bilirubin level and other cholestatic parameters does not occur immediately after SEMS placement.

1.2 Secondary endpoints

* Health-related quality of life (HRQL) (evaluated monthly)
* Complications (perforation, haemorrhage, pancreatitis, cholecystitis, cholangitis, stent migration [into the duodenal lumen by ≥ 1 cm], sludge occlusion, severe pain, tumor in- and over-growth, infection, haemorrhage, stent fracture and shearing, stent cover disruption) major and minor.
* Overall survival post stent placement
* Quality adjusted life years (QALYs)
* Costs of treatment strategies
* Occurrence of biliary re-intervention, defined as any endoscopic, percutaneous or surgical procedure to improve biliary drainage after the stent placement
* Procedure time (stent deployment)
* Technical complications of the tested endoscopic devices. Population: The study population will include patients with symptoms (jaundice, cholangitis) due to malignant extrahepatic biliary tree obstruction (pancreatic cancer, cholangiocarcinoma, gallbladder cancer, or metastatic lymphadenopathy) who are not candidates for surgical cure either because the tumor is inoperable or because of the patient's poor medical condition due to comorbidities and/or advanced age.

Patients with extrahepatic malignancy in whom a diagnostic work up is still ongoing to establish the possibility of performing a curative approach will not be immediately enrolled. Patients who have been previously treated with a plastic stent will be eligible if the plastic stent was placed within the 4 weeks prior to enrolment in this study.

Materials Fully covered SEMS: Niti-S Biliary ComVi Stent; Uncovered SEMS: Niti-S (D type) stent Sample size calculation: The primary end point of the study is stent occlusion. The number of patients in each group required to demonstrate a statistically significant difference in SEMS patency with an 80% power is 70 for a 22% difference,121 for a 17% difference, and 248 for a 12% difference in the obstruction rate between the two groups. Estimated sample size is 121 for a 17% difference, and 70 for a 22% difference.

With a lower (75%) power, 63 patients per treatment group are required to detect a difference of 22%, 108 for a 17% difference and 222 for a 12% difference. This computation is based on data on obstruction percentage reported in literature.

The target enrolment for this study will be 70 patients per study arm. Considering time to occlusion analysis, a total of 140 patients will detect a treatment difference at a two sided 0.05 significance level, with 80% power, if the true hazard ratio is at least 1.76.

Treatment of data Data storage, management, and analysis will be centralized. An electronic database will be constructed to collect the data. The program will be distributed to all participating centers and the data will be entered at the time of the encounters with the subjects such as at the time of endoscopy for stent placement, follow-up visit, or follow-up telephone call. Randomization assignment (stent type) will be coded. Standard operating procedures for regularly backing up the data will be employed at each facility and centrally.

Every 6 months the compact disk (CD) with the study site data will be sent to the coordinating center where the data manger will download the data and merge it with the previously collected study data.

Security measures will be adopted before the mailing of the CD in order to avoid any possible disclosure of the privacy: the data will be encrypted and transformed in numbers.

The data manager will remove information regarding the type of SEMS used prior to sending the data to the statistician. Therefore, data analysis will be performed by a statistician who is blinded to the type of stent.

Data sheet

* Baseline and enrolment visit (Day 0)
* Follow-up visits (1 week, 1 month, 3 and 6 months after stent placement)
* Specific Exams/Tests required Stent placement procedure (Day 0) The patients who agree to participate and who sign a Patient Consent will be enrolled in the study; prior to enrolment, the investigator will provide thorough explanation of the study procedures.

Clinical data (Form A):

* patient demographics (gender, age)
* medical history related to diagnosis and history
* concomitant medications and treatments
* endoscopic and/or MRI and/or CT-scan exam for confirmation and location of stent
* stenosis (the endoscopic examination could be done immediately before the stent placement procedure)
* liver function tests

  1 week, 1 month, 3 and 6 months after placement (Form B):
* liver function tests
* concomitant medications and treatment
* confirmation of stent position via supine X-ray
* Complications 1. week, 1 month, 3 and 6 months after placement (Form E): HRQL questionnaires Analysis Descriptive statistics, including graphical displays, will be used to summarize all study variables. The unit of analysis will be the patient. For continuous variables, means, medians, standard deviations, percentiles, ranges, box plots and histograms will be generated. For categorical variables, frequencies and proportions will be generated. The investigators will examine all variables to determine if parametric distributional assumptions (e.g. normality for the continuous variables) are valid.

Differences between continuous variables will be determined by parametric tests, or, when appropriate by non-parametric tests. Differing frequencies of variables at different times within each group (dysphagia score, body weight, etc) will be compared with tests for related samples.

To address the primary aim, differences in duration of stent patency, the Kaplan-Meier method will be used to estimate stent patency in each group and the log-rank test will be used for an unadjusted comparison between groups. Then a Cox proportional hazard model will be constructed to compare time to stent occlusion adjusted for important potential confounders. Stent patency will be calculated in days and will represent the interval between the time of stent insertion and the time of its replacement or the death of the patient with concomitant cholangitis.

To address the secondary aims, relationships between complication rates and stent type will be examined by the chi-square or the exact Fisher tests. Logistic regression will be used to compare stent complication rates adjusted for important potential confounders. Health-related quality of life (HRQL) will be evaluated by a paired t-test to determine the impact of stent placement (i.e. compare baseline HRQL and month 3 HRQL) by Student's t -test to compare the differences in HRQL at baseline and 3 months between study groups. Linear regression models will be constructed to assess HQRL while adjusting for factors other than stent type. Total direct costs for each study group will be compared and cost effectiveness modelled.

For all analyses the Statistical Package for Social Sciences software (SPSS, Inc. for Windows will be used.

Adverse events are defined as any undesirable experience occurring to a subject during a clinical trial. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded.

A serious adverse event is any untoward medical occurrence or effect that at any level results in death:

* is life threatening (at the time of the event)
* requires hospitalisation or prolongation of existing in patients' hospitalisation
* results in persistent or significant disability or incapacity
* is a new event of the trial likely to affect the safety of the subjects, such as an unexpected outcome of an adverse reaction, lack of efficacy, major safety finding Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Malignant obstructive disease at the level of the extrahepatic bile duct (CBD)
* Serum bilirubin >50 micromol/L
* Inoperability due to a poor medical condition and/or unresectable disease
* ≥ 18 years of age
* Willing and able to comply with study procedures and provide written informed consent

Exclusion Criteria:

* Benign obstruction of the CBD
* Malignancy involving intrahepatic ducts or duodenum
* Prior gastric bypass or Billroth type I or type II gastric resection
* Prior biliary surgery
* World Health Organization (WHO) performance score of 4 (100% of time in bed)
* international normalized ratio (INR)> 1.5
* Life expectancy of < 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To compare the duration of stent patency of a covered vs. an uncovered biliary SEMS placed to relieve biliary obstruction in patients with inoperable extrahepatic malignant biliary obstruction. | minimum follow-up: 4 months
  The Kaplan-Meier method will be used to estimate stent patency in each group and the log-rank test will be used for an unadjusted comparison between groups. Then a Cox proportional hazard model will be constructed to compare time to stent occlusion adjusted for important potential confounders. Stent patency will be calculated in days and will represent the interval between the time of stent insertion and the time of its replacement or the death of the patient with concomitant cholangitis.
To evaluate complication rates of covered vs. uncovered biliary SEMS in patients with inoperable extrahepatic malignant biliary obstruction | minimum follow-up: 4 months
  Relationships between complication rates and stent type will be examined by the chi-square or the exact Fisher tests. Logistic regression will be used to compare stent complication rates adjusted for important potential confounders.

SECONDARY OUTCOMES:
To evaluate the quality of life before and after intervention with covered vs. uncovered biliary SEMS in patients with inoperable extrahepatic malignant biliary obstruction. | 3 months
  Health-related quality of life (HRQL) will be evaluated by a paired t-test to determine the impact of stent placement (i.e. compare baseline HRQL and month 3 HRQL) by Student's t -test to compare the differences in HRQL at baseline and 3 months between study groups. Linear regression models will be constructed to assess HQRL while adjusting for factors other than stent type.
To evaluate the survival of patients treated with covered vs. uncovered biliary SEMS for the management of inoperable extrahepatic malignant biliary obstruction. | until death
  For all analyses the Statistical Package for Social Sciences software (SPSS, Inc. for Windows will be used.
To evaluate the cost-effectiveness of covered and uncovered biliary SEMS in patients with inoperable extrahepatic malignant biliary obstruction | until death
  Total direct costs for each study group will be compared and cost effectiveness modelled.
  For all analyses the Statistical Package for Social Sciences software (SPSS, Inc. for Windows) will be used.
To determine the predictors of survival in patients in patients with inoperable extrahepatic malignant biliary obstruction managed with SEMS. | minimum follow-up: 4 months
  For all analyses the Statistical Package for Social Sciences software (SPSS, Inc. for Windows will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Conio, MD, Principal Investigator — General Hospital Sanremo, Sanremo, Italy
Locations (1):
- General Hospital sanremo, Sanremo, Imperia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warshaw AL, Fernandez-del Castillo C. Pancreatic carcinoma. N Engl J Med. 1992 Feb 13;326(7):455-65. doi: 10.1056/NEJM199202133260706. No abstract available. PMID 1732772
- [Background] Cubiella J, Castells A, Fondevila C, Sans M, Sabater L, Navarro S, Fernandez-Cruz L. Prognostic factors in nonresectable pancreatic adenocarcinoma: a rationale to design therapeutic trials. Am J Gastroenterol. 1999 May;94(5):1271-8. doi: 10.1111/j.1572-0241.1999.01018.x. PMID 10235206
- [Background] Dumonceau JM, Cremer M, Auroux J, Delhaye M, Deviere J. A comparison of Ultraflex Diamond stents and Wallstents for palliation of distal malignant biliary strictures. Am J Gastroenterol. 2000 Mar;95(3):670-6. doi: 10.1111/j.1572-0241.2000.01844.x. PMID 10710055
- [Background] Ferlitsch A, Oesterreicher C, Dumonceau JM, Deviere J, Leban T, Born P, Rosch T, Suter W, Binek J, Meyenberger C, Mullner M, Schneider B, Schofl R. Diamond stents for palliation of malignant bile duct obstruction: a prospective multicenter evaluation. Endoscopy. 2001 Aug;33(8):645-50. doi: 10.1055/s-2001-16214. PMID 11490378
- [Background] Ahmad J, Siqueira E, Martin J, Slivka A. Effectiveness of the Ultraflex Diamond stent for the palliation of malignant biliary obstruction. Endoscopy. 2002 Oct;34(10):793-6. doi: 10.1055/s-2002-34269. PMID 12244500
- [Background] Shah RJ, Howell DA, Desilets DJ, Sheth SG, Parsons WG, Okolo P 3rd, Lehman GA, Sherman S, Baillie J, Branch MS, Pleskow D, Chuttani R, Bosco JJ. Multicenter randomized trial of the spiral Z-stent compared with the Wallstent for malignant biliary obstruction. Gastrointest Endosc. 2003 Jun;57(7):830-6. doi: 10.1016/s0016-5107(03)70016-9. PMID 12776028
- [Background] Kaassis M, Boyer J, Dumas R, Ponchon T, Coumaros D, Delcenserie R, Canard JM, Fritsch J, Rey JF, Burtin P. Plastic or metal stents for malignant stricture of the common bile duct? Results of a randomized prospective study. Gastrointest Endosc. 2003 Feb;57(2):178-82. doi: 10.1067/mge.2003.66. PMID 12556780
- [Background] Knyrim K, Wagner HJ, Pausch J, Vakil N. A prospective, randomized, controlled trial of metal stents for malignant obstruction of the common bile duct. Endoscopy. 1993 Mar;25(3):207-12. doi: 10.1055/s-2007-1010294. PMID 8519239
- [Background] Saito H, Sakurai Y, Takamura A, Horio K. [Biliary endoprosthesis using Gore-Tex covered expandable metallic stents: preliminary clinical evaluation]. Nihon Igaku Hoshasen Gakkai Zasshi. 1994 Feb 25;54(2):180-2. Japanese. PMID 8121783
- [Background] Isayama H, Komatsu Y, Tsujino T, Sasahira N, Hirano K, Toda N, Nakai Y, Yamamoto N, Tada M, Yoshida H, Shiratori Y, Kawabe T, Omata M. A prospective randomised study of "covered" versus "uncovered" diamond stents for the management of distal malignant biliary obstruction. Gut. 2004 May;53(5):729-34. doi: 10.1136/gut.2003.018945. PMID 15082593
- [Background] Park DH, Kim MH, Choi JS, Lee SS, Seo DW, Kim JH, Han J, Kim JC, Choi EK, Lee SK. Covered versus uncovered wallstent for malignant extrahepatic biliary obstruction: a cohort comparative analysis. Clin Gastroenterol Hepatol. 2006 Jun;4(6):790-6. doi: 10.1016/j.cgh.2006.03.032. Epub 2006 May 22. PMID 16716757
- [Background] Yoon WJ, Lee JK, Lee KH, Lee WJ, Ryu JK, Kim YT, Yoon YB. A comparison of covered and uncovered Wallstents for the management of distal malignant biliary obstruction. Gastrointest Endosc. 2006 Jun;63(7):996-1000. doi: 10.1016/j.gie.2005.11.054. PMID 16733115
- [Background] Isayama H, Kawabe T, Nakai Y, Tsujino T, Sasahira N, Yamamoto N, Arizumi T, Togawa O, Matsubara S, Ito Y, Sasaki T, Hirano K, Toda N, Komatsu Y, Tada M, Yoshida H, Omata M. Cholecystitis after metallic stent placement in patients with malignant distal biliary obstruction. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1148-53. doi: 10.1016/j.cgh.2006.06.004. Epub 2006 Aug 14. PMID 16904950
- [Background] Davids PH, Groen AK, Rauws EA, Tytgat GN, Huibregtse K. Randomised trial of self-expanding metal stents versus polyethylene stents for distal malignant biliary obstruction. Lancet. 1992 Dec 19-26;340(8834-8835):1488-92. doi: 10.1016/0140-6736(92)92752-2. PMID 1281903
- [Background] Prat F, Chapat O, Ducot B, Ponchon T, Pelletier G, Fritsch J, Choury AD, Buffet C. A randomized trial of endoscopic drainage methods for inoperable malignant strictures of the common bile duct. Gastrointest Endosc. 1998 Jan;47(1):1-7. doi: 10.1016/s0016-5107(98)70291-3. PMID 9468416